CLINICAL TRIAL: NCT05290571
Title: The Effectiveness of Modified Otago Exercise Program on Balance Performance of Elderlies in Hong Kong
Brief Title: Modified Otago Exercise Program on Balance Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Ho Yuk Ki Yorke, Student physiotherapist, Tung Wah College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHS_SRC_2021_001
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Healthy Aging; Fall
Keywords: Modified Otago Exercise Program; Modified Otago Exercise Program with music

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group will be asked to follow the actions in the provided video. It lasts for approximately 30 minutes, with 5-minute warm-up and cool-down exercises respectively, a 4-minute song repeating for 4 times and a 1-minute rest in between each repetition. Videos, in the form of a YouTube link, will be distributed for the Intervention Group, as well as the leaflets.
  Interventions: Other: Modified Otago Exercise Program with music
- Control Group (Active Comparator): Control Group will receive a leaflet on 10 actions extracted from mOEP, 2 actions from conventional OEP and 1 action from Mini-BESTest. The participants will perform 8-16 repetitions for each action, with 3-5 seconds of rest between actions.
  Interventions: Other: Modified Otago Exercise Program

INTERVENTIONS:
Other: Modified Otago Exercise Program with music — Our study attempts to establish a new home-based exercise option incorporating mOEP with video, music and lyrics. Our new approach shares the same aims with Exergames and video-supported methods - to increase the exercise motivation of elderlies, hence their physical performance. Based on the video-supported approach in one previous study, we add in the component of music therapy. Music-based exercise interventions could produce positive outcomes on both physical, such as gait, balance and fall risk and level of physical activities and psychological, including exercise adherence, perceived exertion, thus extending exercise duration. However, exact mechanisms have not been revealed and it may be limited by personal preferences on music. In our video, the music we chose is of brisk rhythm, slightly delightful melody and higher pitch, which all help to shape a cheerful and relaxing atmosphere for the elderlies.
  Arms: Intervention Group
Other: Modified Otago Exercise Program — Otago Exercise Program (OEP) was developed by Otago Medical School in New Zealand as a tailor-made home-based fall prevention program to improve the balance performance of community-dwelling elderlies over 1 year. It comprises of 3 main components: 5 lower limb strengthening, 12 balance retraining and walking exercises. In the original program, the intensity was set as moderate with up to 4 difficulty levels for strengthening and balance exercises, in terms of ankle cuff weights and number of repetitions, and level of support respectively. It also stated that the frequency was at least 3 times a week for the former two exercises and at least 2 times per week for walking exercises; while the total duration was expected to make up to an hour, including 30-minute walking exercises.
  Arms: Control Group

SUMMARY:
Fall is a common problem encountered by elderlies. In Hong Kong, the prevalence rate of falls among elderlies aged above 65 years old ranged from 18%-29%, standing at approximately one-fifths of the total elderly population. Falls pose huge threats to the physical and psychosocial health of the elderlies as they are often accompanied by serious injuries such as bone fracture and post-fall syndrome, decreased confidence in walking, and social exclusion.

Otago Exercise Program (OEP) was a tailor-made home-based fall prevention program of community-dwelling elderlies. It comprises of 3 main components: 5 lower limb strengthening, 12 balance retraining and walking exercises. Regarding on its effectiveness, multiple studies revealed that OEP and modified version of OEP (mOEP) brought significant improvements on perceived, static and dynamic balance, lower limb strength, quality of life and functional capacity of healthy elderlies and those with various health conditions such as chronic illnesses, osteoarthritis, stroke and hemiplegia.

The delivery method of OEP and mOEP has been limited to have elderlies following the instructions and illustrations of a printed booklet. Currently, there are only two proposed effective forms of mOEP: video-instructed and Exergames. Our study attempts to establish a new home-based exercise option incorporating mOEP with video, music and lyrics. It helps to increase the exercise motivation of elderlies, hence their physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Elderlies in community dwellings aged 55 or above
* Communicable & able to follow command
* Self-reported sufficient visual & auditory ability to follow the actions in video
* HK-MoCA 5-Min Protocol: No cognitive impairment
* Able to access electronic devices, such as smartphones, computers, televisions with network, Digital Video Disc/Compact Disc player

Exclusion Criteria:

* History of severe medical conditions that hinders physical ability, such as heart diseases and neurological disorders
* History of lower limb fracture in recent 1 year
* History of joint replacement and any cardio-thoracic surgeries
* Self-reported visual & auditory impairment
* Users of walking aids other than sticks, tripods or quadripods

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Falls Efficacy Scale International (FES-I) | 1 week before the Intervention
  The Falls Efficacy Scale-International (FES-I) is a modified version of the FES, based on the perceptive feeling on fall risks of the participants. It is a 16-item questionnaire on a 4-point ordinal scale, emphasizing social and physical activities. The minimum and maximum score is 16 and 64 respectively while a lower score indicates higher confidence in one's balance ability.
Falls Efficacy Scale International (FES-I) | 4 weeks after the start of the Intervention
Falls Efficacy Scale International (FES-I) | 1 week after the completion of the Intervention
Change from Falls Efficacy Scale International (FES-I) at 4 weeks | 1 week before the Intervention, 4 weeks after the start of the Intervention
Change from Falls Efficacy Scale International (FES-I) at 8 weeks | 1 week before the Intervention, 1 week after the completion of the Intervention
Change of Falls Efficacy Scale International (FES-I) between 4 weeks and 8 weeks | 4 weeks after the start of the Intervention, 1 week after the completion of the Intervention
Functional Reach Test (FRT) | 1 week before the Intervention
  Functional Reach Test (FRT) is a common clinical outcome measure on dynamic standing balance. The participants were required to stand adjacent to a wall with a meter ruler fixed and to raise their preferred upper limb to the shoulder level. They were then instructed to reach as far as possible while maintaining their balance without moving both lower limbs for two trials, following one mock trial. The result recorded was the average distance from the reading of the tip of the third digit of the two trials. The longer the subject reaches, the better their dynamic balance.
Functional Reach Test (FRT) | 4 weeks after the start of the Intervention
Functional Reach Test (FRT) | 1 week after the completion of the Intervention
Change from Functional Reach Test (FRT) at 4 weeks | 1 week before the Intervention, 4 weeks after the start of the Intervention
Change from Functional Reach Test (FRT) at 8 weeks | 1 week before the Intervention, 1 week after the completion of the Intervention
Change of Functional Reach Test (FRT) between 4 weeks and 8 weeks | 4 weeks after the start of the Intervention, 1 week after the completion of the Intervention
Mini Balance Evaluation Systems Test (Mini-BESTest) | 1 week before the Intervention
  The Mini Balance Evaluation Systems Tests (Mini-BESTest) emphasizes on measuring dynamic balance, functional mobility and gait. The total score is 28 and encompasses 14 items, including anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. Subjects were asked to perform 14 actions such as sit to stand, tip-toe standing and single leg standing. A higher score indicates better balance ability of the subjects.
Mini Balance Evaluation Systems Test (Mini-BESTest) | 4 weeks after the start of the Intervention
Mini Balance Evaluation Systems Test (Mini-BESTest) | 1 week after the completion of the Intervention
Changes from Mini Balance Evaluation Systems Test (Mini-BESTest) at 4 weeks | 1 week before the Intervention, 4 weeks after the start of the Intervention
Changes from Mini Balance Evaluation Systems Test (Mini-BESTest) at 8 weeks | 1 week before the Intervention, 1 week after the completion of the Intervention
Changes of Mini Balance Evaluation Systems Test (Mini-BESTest) between 4 weeks and 8 weeks | 4 weeks after the start of the Intervention, 1 week after the completion of the Intervention

SECONDARY OUTCOMES:
Montreal Cognitive Assessment 5-minute protocol (Hong Kong version (HK-MoCA 5-min protocol) | 1 week before the Intervention
  The Montreal Cognitive Assessment 5-minute protocol (MoCA 5-min protocol) version 20151030 is an abbreviated Chinese version of conventional MoCA, including 4 subtests. It emphasizes on the examination of 5 cognitive domains, which incorporates attention, verbal learning and memory, executive function and orientation. Participants were required to recall 5 words from the first trial, name animals for 1 minute, answer 6 items on date and geographic orientation and to remember the 5 words provided at the beginning of the test. The maximum score for the test is 30 while a higher outcome indicates better cognitive ability.
Montreal Cognitive Assessment 5-minute protocol (Hong Kong version (HK-MoCA 5-min protocol) | 4 weeks after the start of the Intervention
Montreal Cognitive Assessment 5-minute protocol (Hong Kong version (HK-MoCA 5-min protocol) | 1 week after the completion of the Intervention
Changes from Montreal Cognitive Assessment 5-minute protocol (Hong Kong version (HK-MoCA 5-min protocol) at 4 weeks | 1 week before the Intervention, 4 weeks after the start of the Intervention
Changes from Montreal Cognitive Assessment 5-minute protocol (Hong Kong version (HK-MoCA 5-min protocol) at 8 weeks | 1 week before the Intervention, 1 week after the completion of the Intervention
Changes of Montreal Cognitive Assessment 5-minute protocol (Hong Kong version (HK-MoCA 5-min protocol) between 4 weeks and 8 weeks | 4 weeks after the start of the Intervention, 1 week after the completion of the Intervention
Physical Activity Scale for the Elderly - Chinese version (PASE-C) | 1 week before the Intervention
  The Physical Activity Scale for the Elderly - Chinese version (PASE-C) is a brief assessment on the usual physical activity of the elderlies over a week. PASE scores are divided into three categories: sedentary, light, and moderate to intense. It examines the intensity of participation in leisure activities, sports, recreation, and muscle strengthening, and work. A higher score means that the subject adopts a more active lifestyle.
Physical Activity Scale for the Elderly - Chinese version (PASE-C) | 4 weeks after the start of the Intervention
Physical Activity Scale for the Elderly - Chinese version (PASE-C) | 1 week after the completion of the Intervention
Changes from Physical Activity Scale for the Elderly - Chinese version (PASE-C) at 4 weeks | 1 week before the Intervention, 4 weeks after the start of the Intervention
Changes from Physical Activity Scale for the Elderly - Chinese version (PASE-C) at 8 weeks | 1 week before the Intervention, 1 week after the completion of the Intervention
Changes of Physical Activity Scale for the Elderly - Chinese version (PASE-C) between 4 weeks and 8 weeks | 4 weeks after the start of the Intervention, 1 week after the completion of the Intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Tung Wah College, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhambra-Borrás, T., Valia-Cotanda, E., Dura-Ferrandis, E., Garcés-Ferrer, J. & Quel-Tejón, B. (2017). Promoting active ageing through a physical exercise program aimed at reducing frailty and risk of failing among older adults. International Journal of Integrated Care, 17(5): A225, 1-8. Doi: dx.doi.org/10.5334/ijic.3535.
- [Background] Almarzouki R, Bains G, Lohman E, Bradley B, Nelson T, Alqabbani S, Alonazi A, Daher N. Improved balance in middle-aged adults after 8 weeks of a modified version of Otago Exercise Program: A randomized controlled trial. PLoS One. 2020 Jul 15;15(7):e0235734. doi: 10.1371/journal.pone.0235734. eCollection 2020. PMID 32667956
- [Background] Campbell, A.J. & Robertson, M.C. (2003). Otago Exercise Programme to prevent falls in older adults. Otago Medical School. Retrieved from https://www.livestronger.org.nz/assets/Uploads/acc1162-otago-exercise-manual.pdf
- [Background] Chiu HL, Yeh TT, Lo YT, Liang PJ, Lee SC. The effects of the Otago Exercise Programme on actual and perceived balance in older adults: A meta-analysis. PLoS One. 2021 Aug 6;16(8):e0255780. doi: 10.1371/journal.pone.0255780. eCollection 2021. PMID 34358276
- [Background] Chu, L.W., Chi, I. & Chiu, A.Y.Y. (2007). Falls and fall-related injuries in community-dwelling elderly persons in Hong Kong: a study on risk factors, functional decline, and health services utilization after falls. Hong Kong Medical Journal. 2007; 13(Suppl 1): S8-12. Retrieved from https://www.hkmj.org/system/files/hkm0702sp1p8.pdf
- [Background] Dadgari A, Aizan Hamid T, Hakim MN, Chaman R, Mousavi SA, Poh Hin L, Dadvar L. Randomized Control Trials on Otago Exercise Program (OEP) to Reduce Falls Among Elderly Community Dwellers in Shahroud, Iran. Iran Red Crescent Med J. 2016 Feb 14;18(5):e26340. doi: 10.5812/ircmj.26340. eCollection 2016 May. PMID 27478629
- [Background] Department of Health. (2019). Fall Prevention in Elderly. Elderly Health Service of Department of Health and Primary Healthcare Office of Food and Health Bureau. Retrieved from https://www.elderly.gov.hk/tc_chi/books/files/fall_prevention/Fall_Prevention_booklet.pdf
- [Background] Fong, K.N.K., Siu, A.M.H., Au Yeung, K., Cheung, S.W.S. & Chan, C.C.H. (2011). Falls among the Community-living elderly people in Hong Kong: A retrospective study. Hong Kong Journal of Occupational Therapy. 21; 1: 33-40. Doi: 10.106/j.hkjot.2011.05.005.
- [Background] Jose, S. & Sangita, K. (2018). Effectiveness of Otago exercise to improve balance, quality of life and to reduce risk of fall in hemiplegic patients. International Journal of Science and Research (IJSR). 2019, Vol. 8, (8), 2043-46. Retrieved from https://www.ijsr.net/archive/v8i8/ART2020776.pdf
- [Background] Kiik, S.M., Vanchapo, A.R., Elfrida, M.F., Nuwa, M.S. & Sakinah, S. (2020). Effectiveness of Otago exercise on health status and risk of fall among elderly with chronic illness. Jurnal Keperawatan Indonesia. 2020; 23 (1), 15-22. Doi: 10.7454/jki.v23il.900.
- [Background] Luk JK, Chan TY, Chan DK. Falls prevention in the elderly: translating evidence into practice. Hong Kong Med J. 2015 Apr;21(2):165-71. doi: 10.12809/hkmj144469. Epub 2015 Feb 27. PMID 25722468
- [Background] Martins AC, Guia D, Saraiva M, Pereira T. Effects of A "Modified" Otago Exercise Program on the Functional Abilities and Social Participation of Older Adults Living in the Community-The AGA@4life Model. Int J Environ Res Public Health. 2020 Feb 15;17(4):1258. doi: 10.3390/ijerph17041258. PMID 32075307
- [Background] Park Y, Chang M. Effects of the Otago exercise program on fall efficacy, activities of daily living and quality of life in elderly stroke patients. J Phys Ther Sci. 2016 Jan;28(1):190-3. doi: 10.1589/jpts.28.190. Epub 2016 Jan 30. PMID 26957755
- [Background] Salekar, S. & Khandale, S.R. (2019). Effect of Otago exercise program on balance and risk of fall in community-dwelling individuals having knee osteoarthritis. International Journal of Advance Research and Development. Vol. 4, (4): 36-38. Retrieved from https://www.ijarnd.com/manuscripts/v4i4/V4I4-1152.pdf
- [Background] Stanmore EK, Mavroeidi A, de Jong LD, Skelton DA, Sutton CJ, Benedetto V, Munford LA, Meekes W, Bell V, Todd C. The effectiveness and cost-effectiveness of strength and balance Exergames to reduce falls risk for people aged 55 years and older in UK assisted living facilities: a multi-centre, cluster randomised controlled trial. BMC Med. 2019 Feb 28;17(1):49. doi: 10.1186/s12916-019-1278-9. PMID 30813926
- [Background] Benavent-Caballer V, Rosado-Calatayud P, Segura-Orti E, Amer-Cuenca JJ, Lison JF. The effectiveness of a video-supported group-based Otago exercise programme on physical performance in community-dwelling older adults: a preliminary study. Physiotherapy. 2016 Sep;102(3):280-6. doi: 10.1016/j.physio.2015.08.002. Epub 2015 Sep 1. PMID 26395209